CLINICAL TRIAL: NCT06044337
Title: A Multicenter, Open-Label, Single-Arm, Phase 3, Long-Term Extension Study to Evaluate Continuous Safety and Efficacy of BIIB059 (Litifilimab) in Adult Participants With Active Subacute Cutaneous Lupus Erythematosus and/or Chronic Cutaneous Lupus Erythematosus With or Without Systemic Manifestations and Refractory and/or Intolerant to Antimalarial Therapy
Brief Title: A Long-Term Extension Study to Learn More About the Safety of Litifilimab (BIIB059) Injections and Whether They Can Improve Symptoms of Adult Participants Who Have Active Cutaneous Lupus Erythematosus
Acronym: AMETHYST LTE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230LE305; 2023-504863-17-00 (Other: EU CTIS Number)
Record Dates: First submitted 2023-08-23; First posted 2023-09-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Subacute Cutaneous Lupus Erythematosus; Chronic Cutaneous Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BIIB059 (Experimental): Participants will receive BIIB059 (litifilimab) subcutaneously (SC), once every 4 weeks up to Week 100 in the LTE period. Following the 2 year long-term extension (LTE) period, participants in the USA will receive BIIB059 (litifilimab), once every 4 weeks up to Week 256.
  Interventions: Drug: BIIB059 (litifilimab)

INTERVENTIONS:
Drug: BIIB059 (litifilimab) — Administered as specified in the treatment arm.
  Other Names: litifilimab

SUMMARY:
In this study, researchers will learn more about a study drug called BIIB059 (litifilimab) in participants with cutaneous lupus erythematosus (CLE). The study will focus on participants who have either active subacute CLE or chronic CLE, or both. They may also have systemic lupus erythematosus (SLE). The participants did not respond to antimalarial therapy or had problems with the treatment that made it hard to continue.

The study will enroll only those participants who have completed treatment with litifilimab in the parent study, 230LE301.

The main objective of the study is to learn more about the long-term safety of litifilimab.

The main question researchers want to answer is:

- How many participants have adverse events and serious adverse events after taking litifilimab? Adverse events are unwanted health problems that may or may not be caused by the study drug.

Researchers will also learn more about the effect of litifilimab on CLE. They will do this by measuring the symptoms of CLE over time using a variety of scoring tools. These include the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI), the Cutaneous Lupus Activity of Investigator's Global Assessment-Revised (CLA-IGA-R), and the SELENA-SLEDAI Flare Index (SFI).

Researchers will look at how litifilimab and CLE affect the quality of life of participants using a group of questionnaires. They will also look at how litifilimab affects laboratory tests and how participants' immune systems respond to litifilimab.

The study will be done as follows:

* The last visit of parent study 230LE301 will be the first visit of study 230LE305.
* All participants will receive litifilimab as an injection under the skin once every 4 weeks. Both researchers and participants will know the dose and identity of the study drug.
* Globally, the treatment period will last up to 104 weeks, or 2 years. For participants in the United States, the treatment period may last up to 260 weeks, or 5 years
* There will be a follow-up safety period that lasts up to 24 weeks.
* Globally, participants will have up to 27 study visits during the treatment period. In the US, participants will have up to 66 study visits.
* Globally, the total study duration for participants will be up to 128 weeks. In the US, the total study duration will be up to 284 weeks .

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the long-term safety and tolerability BIIB059 (litifilimab) in participants who completed the parent study 230LE301 (NCT05531565) with active subacute CLE and/or chronic CLE with or without systemic manifestations and refractory and/or intolerant to antimalarial therapy.

The secondary objectives of the study are to evaluate the long-term effect of litifilimab on disease activity and the effect of litifilimab in preventing disease damage in participants with active subacute CLE and/or chronic CLE with or without systemic manifestations and refractory and/or intolerant to antimalarials; to evaluate the long-term effect of litifilimab on preventing lupus flare in participants with CLE with SLE; to assess long-term use of oral corticosteroid (OCS) in participants receiving litifilimab treatment; to assess the impact of litifilimab on participant-reported health-related quality of life (HRQoL); to evaluate long-term effect of litifilimab on laboratory parameters; to evaluate the immunogenicity and pharmacokinetics (PK) of litifilimab.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who completed the parent study (230LE301 [NCT05531565], Part A or Part B) on study treatment (received treatment through Week 48 and attended the last study assessment visit at Week 52).
* Ability of the participant to understand the purpose and risks of the study, to provide informed consent, and to authorize the use of confidential health information in accordance with national and local privacy regulations.

Key Exclusion Criteria:

* Early Part A or Part B parent study (230LE301 [NCT05531565]) treatment terminators (participants who discontinued study treatment before Week 48).
* Early Part A or Part B parent study terminators [participants who withdrew from parent study participation before Week 52 and did not complete the parent study extended treatment period (ETP)].
* Participants who have developed any other medical diseases, conditions, or abnormalities, rendering their participation in the long-term extension (LTE) study unsuitable in the opinion of the Investigator.

NOTE: Other protocol- defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2029-06-26 (Estimated); Study Completion 2029-12-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 128 weeks

SECONDARY OUTCOMES:
Percentage of Participants who Achieve a Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity Score (CLASI)-70 Response, Defined as a 70% Improvement in CLASI-A Score From the Baseline Value (Parent Study [NCT05531565]) | Up to 128 weeks
Percentage of Participants who Achieve a CLASI-50 Response, Defined as a 50% Improvement in CLASI-A Score From the Baseline Value (Parent Study [NCT05531565]) | Up to 128 weeks
Percentage of Participants who Achieve a CLASI-90 Response, Defined as a 90% Improvement in CLASI-A Score From the Baseline Value (Parent Study [NCT05531565]) | Up to 128 weeks
Percentage of Participants who Achieve a Cutaneous Lupus Activity of Physician's Global Assessment-Revised (CLA-IGA-R) Erythema Score of 0 or 1 | Up to 128 weeks
Percentage of Participants who Achieve a CLA-IGA-R Other Morphologic Characteristics (OMC) Score of 0 or 1 | Up to 128 weeks
Cumulative Duration of Sustained CLASI-70 Response, Defined as the Number of Weeks With 70% Improvement in CLASI-A Score From the Baseline Value (Parent Study [NCT05531565]) | Up to 128 weeks
Cumulative Duration of Sustained CLASI-50 Response, Defined as the Number of Weeks With 50% Improvement in CLASI-A Score From the Baseline Value (Parent Study [NCT05531565]) | Up to 128 weeks
Cumulative Duration of Sustained CLASI-90 Response, Defined as the Number of Weeks With 90% Improvement in CLASI-A Score From the Baseline Value (Parent Study [NCT05531565]) | Up to 128 weeks
Cumulative Duration of Sustained Efficacy, Defined as the Number of Weeks With CLA-IGA-R Erythema Score of 0 or 1 | Up to 128 weeks
Cumulative Duration of Sustained Efficacy, Defined as the Number of Weeks With CLA-IGA-R OMC Score of 0 or 1 and Improvement of at Least 1 Point From Baseline Value (Parent Study [NCT05531565]) | Up to 128 weeks
Cumulative Duration of Sustained Efficacy, Defined as the Number of Weeks With CLA-IGA-R Follicular Activity Score of 0 | Up to 128 weeks
Percentage of Participants With a CLASI-70 Response Among CLASI-70 Responders at Week 52 of the Parent Study (NCT05531565) | Day 0 (Week 52 of parent study) up to 128 weeks
Percentage of Participants With a CLASI-50 Response Among CLASI-50 Responders at Week 52 of the Parent Study (NCT05531565) | Day 0 (Week 52 of parent study) up to 128 weeks
Percentage of Participants With a CLASI-90 Response Among CLASI-90 Responders at Week 52 of the Parent Study (NCT05531565) | Day 0 (Week 52 of parent study) up to 128 weeks
Percentage of Participants With a CLA-IGA-R Erythema Score of 0 or 1 Among Participants With a CLA-IGA-R Erythema Score of 0 or 1 at Week 52 of the Parent Study (NCT05531565) | Day 0 (Week 52 of parent study) up to 128 weeks
Percentage of Participants With CLA-IGA-R OMC Score of 0 or 1 and at Least 1 Level of Improvement From Baseline Value(Parent Study) Among Participants With CLA IGA R OMC Score of 0 or 1 and at Least 1 Level Improvement From Baseline Value(Parent Study) | Day 0 (Week 52 of parent study) up to 128 weeks
Percentage of Participants With a CLASI-70 Response Among CLASI-50 Responders at Week 52 of the Parent Study (NCT05531565) | Day 0 (Week 52 of parent study) up to 128 weeks
Percentage of Participants With a CLASI-90 Response Among CLASI-50 Responders at Week 52 of the Parent Study (NCT05531565) | Day 0 (Week 52 of parent study) up to 128 weeks
Percentage of Participants With a CLASI-90 Response Among CLASI-70 Responders at Week 52 of the Parent Study (NCT05531565) | Day 0 (Week 52 of parent study) up to 128 weeks
Percentage of Participants With Loss of Response, Defined as an Increase of ≥ 7 Points in CLASI-A Total Score From Baseline | Baseline (Day 0) up to 128 weeks
Percentage of Participants With Loss of Response, Defined as Achieving 2 Points Improvement From Baseline Value(Parent Study) CLA-IGA-R Erythema Score at Beginning of/During LTE Study and Then Relapsing to CLA-IGA-R Erythema Baseline Value(Parent Study) | Up to 128 weeks
Percentage of Participants With Loss of Response, Defined as Having at Least 2, 3, and 4 Points Worsening in CLA-IGA-R Erythema Score From Their Minimum Score in the Parent Study (NCT05531565) | Up to 128 weeks
Absolute Change in Cutaneous Lupus Erythematosus Disease Area and Severity Index Damage (CLASI-D) Score From Baseline Value (Parent Study [NCT05531565]) to Week 104 | Up to 104 weeks
Percent Change in CLASI-D Score From Baseline Value (Parent Study [NCT05531565]) to Week 104 | Up to 104 weeks
Annualized Mild/Moderate and Severe Safety of Estrogens in Lupus Erythematosus National Assessment-SLE Disease Activity Index Flare Index (SFI) Rates Through Week 52 | Up to 52 weeks
Annualized Mild/Moderate and Severe SFI Rates Through Week 104 | Up to 104 weeks
Percentage of Participants With Oral Corticosteroid (OCS) Dose | Up to 104 weeks
Percentage of Participants With OCS ≤ 7.5 Milligrams per day (mg/day) | Up to 104 weeks
Percentage of Participants With OCS ≤ 5.0 mg/day | Up to 104 weeks
Change From Baseline Value (Parent Study [NCT05531565]) in Cutaneous Lupus Erythematosus - Quality of Life (CLE-QoL) at Weeks 52 and 104 | Baseline, Weeks 52 and 104
Change From Baseline Value (Parent Study [NCT05531565]) in European Quality of Life - 5-Dimensions Questionnaire, 3-Level Version (EQ-5D-3L) at Weeks 52 and 104 | Baseline, Weeks 52 and 104
Change From Baseline Value (Parent Study [NCT05531565]) in 36-Item Short Form Survey (SF-36) (acute version) at Weeks 52 and 104 | Baseline, Weeks 52 and 104
Change From Baseline Value (Parent Study [NCT05531565]) in Work Productivity and Activity Impairment (WPAI): Lupus at Weeks 52 and 104 | Baseline, Weeks 52 and 104
Change From Baseline Value (Parent Study [NCT05531565]) in Patient Health Questionnaire-9 (PHQ-9) at Weeks 52 and 104 | Baseline, Weeks 52 and 104
Change From Baseline Value (Parent Study [NCT05531565]) in Subject Global Assessment of Skin - Follow-up (SGA-Skin-FU) at Weeks 52 and 104 | Baseline, Weeks 52 and 104
Change From Baseline Value (Parent Study [NCT05531565]) in Numerical Rating Scale (NRS) for Pain in Skin Rash at Weeks 52 and 104 | Baseline, Weeks 52 and 104
Change From Baseline Value (Parent Study [NCT05531565]) in Numerical Rating Scale (NRS) for Itch in Skin Rash at Weeks 52 and 104 | Baseline, Weeks 52 and 104
Number of Participants With Clinically Relevant Change From Baseline Value (Parent Study [NCT05531565]) in Standard Laboratory Parameters | Up to 128 weeks
Number of Participants With Clinically Relevant Change From Baseline Value (Parent Study [NCT05531565]) in Electrocardiogram (ECG) Results | Up to 104 weeks
Number of Participants With Anti-BIIB059 Antibodies in Serum | Up to 128 weeks
Serum Concentration of Litifilimab | Pre-dose up to 128 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (86):
- United States (11):
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Dermatology Research Associates, Los Angeles, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - David Fivenson, MD, Dermatology, PLLC, Ann Arbor, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Saint Louis University, St Louis, Missouri
  - Thurston Arthritis Research Center, Chapel Hill, North Carolina
  - Duke Dermatology South Durham, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Precision Comprehensive Clinical Research Solutions, Grapevine, Texas
- Argentina (3):
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - APRILLUS Asistencia e Investigacion, Buenos Aires
- Brazil (6):
  - L2IP - Instituto de Pesquisas Clínicas Ltda., Brasília, Federal District
  - IPC MT Instituto de Pesquisas Clinicas do Mato Grosso, Santo Ângelo, Mato Grosso
  - CMiP - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos, São Paulo, São Paulo
  - IDERJ - Instituto de Dermatologia e Estética do Brasil Ltda, Rio de Janeiro
- Bulgaria (2):
  - DCC 'Alexandrovska', EOOD, Sofia
  - DCC Focus 5 - MEOH OOD, Sofia
- Canada (2):
  - Laser Rejuvenation Clinics, Inc., Calgary, Alberta
  - DIEX Recherche Sherbrooke Inc., Sherbrooke, Quebec
- Chile (3):
  - Centro Medico SkinMed, Las Condes
  - CIEC - Centro Internacional de Estudios Clínicos, Santiago
  - Clinical Research Chile SpA, Valdivia
- China (7):
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Dongguan People's Hospital, Dongguan, Guangdongsheng
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdongsheng
  - The second Xiangya Hospital of Central South University, Changsha, Húnánsheng
  - Hospital for Skin Diseases, Chinese Academy of Medical Sciences, Nanjing, Jiangsu
  - Shanghai Skin Disease Hospital, Shanghai, Shànghaishì
- Colombia (2):
  - Healthy Medical Center, Zipaquirá, Cundinamarca
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
- France (5):
  - CHU de Caen - Hopital de la Cote de Nacre, Caen, Calvados
  - Hopital Larrey, Toulouse, Haute Garonne
  - Hopital Saint Eloi, Montpellier, Herault
  - Hopital Edouard Herriot - CHU Lyon, Lyon, Rhone
  - Hopital Tenon, Paris
- Germany (7):
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Fachklinik Bad Bentheim Dermatologie, Bad Bentheim, Lower Saxony
  - Klinikum Oldenburg AoeR, Oldenburg, Lower Saxony
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus TU, Dresden, Saxony
  - Universitaetsklinikum Halle (Saale), Halle, Saxony-Anhalt
  - Charité - Campus Charité Mitte, Berlin
- Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs, Hungary
- Italy (2):
  - Università degli studi di Firenze, Florence
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
- Japan (11):
  - NHO Nagoya Medical Center, Nagoya, Aichi-ken
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu-shi, Fukuoka
  - Kakogawa Central City Hospital, Kakogawa-shi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Osaka Keisatsu Hospital, Osaka, Osaka
  - Teikyo University Hospital, Itabashi-ku, Tokyo-To
- Mexico (3):
  - Clinstile, S.A. de C.V., Mexico City, Mexico City
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
  - Centro de investigacion medica y reumatologia, Guadalajara
- Philippines (3):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - Lorma Medical Center, San Fernando City, La Union, La Union
  - University of the Philippines Manila - Philippine General Hospital, Manila
- Serbia (2):
  - Institute of Rheumatology_Belgrade, Belgrade
  - University Clinical Center of Serbia, Belgrade
- Artromac n.o., Košice, Slovakia
- South Korea (2):
  - Hanyang University Seoul Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (5):
  - Hospital Universitario Rio Hortega, Valladolid, Cantabria
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
- Karolinska Universitetssjukhuset - Solna, Solna, Sweden
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Lucerne (Luzern)
  - Kantonsspital St. Gallen, Sankt Gallen
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - Whipps Cross University Hospital, London, Greater London
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - Chapel Allerton Hospital, Chapel Allerton, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/